CLINICAL TRIAL: NCT04133935
Title: Prospective Review of Laparoscopic Burch Urethropexy Compared With a Novel Technique of Laparoscopic Obturator Urethropexy: A Randomized Controlled Trial
Brief Title: Treating Stress Urinary Incontinence: Laparoscopic Obturator Urethropexy vs Burch Urethropexy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID restrictions this study has been temporarily halted.
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Nucelio Luiz de Barros Moreira Lemos MD, PhD, Principal Investigator, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0210-A
Record Dates: First submitted 2019-09-30; First posted 2019-10-21 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Upon recruitment to the study, the surgeon will then open a sequentially numbered, opaque, sealed envelope that will randomize the patient to either receiving Burch colposuspension or LOU. The patient will not be made aware of the group they were allocated to.
  A clinical staff who was not involved with the surgery and blinded to the allocation of the patient will complete the Post-operative Follow-up Form at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Obturator Urethropexy (Experimental): Suspending the periurethral vaginal tissue to the obturator internus fascia bilaterally via sutures, creating a support for the bladder neck compartment
  Interventions: Procedure: Laparoscopic Obturator Urethropexy
- Burch Urethropexy (Active Comparator): Suspending the periurethral vaginal tissue to Cooper's ligament bilaterally via sutures, creating a support for the bladder neck compartment
  Interventions: Procedure: Burch Urethropexy

INTERVENTIONS:
Procedure: Laparoscopic Obturator Urethropexy — Suspending the periurethral vaginal tissue to the obturator internus fascia bilaterally via sutures, creating a support for the bladder neck compartment.
  Arms: Laparoscopic Obturator Urethropexy
Procedure: Burch Urethropexy — Suspending the periurethral vaginal tissue to Cooper's ligament bilaterally via sutures, creating a support for the bladder neck compartment
  Arms: Burch Urethropexy

SUMMARY:
Stress urinary incontinence (SUI) is a highly prevalent concern within the female population. Although mid urethral slings (MUS) have been the first line treatment for SUI for almost twenty years, due to recent FDA warnings and many countries banning the use of vaginal mesh, a significant portion of patients now request non-mesh anti-incontinence procedures. In such cases, Burch colposuspension would be the next option discussed with patients.

In the short term, the efficacy of Burch colposuspension is comparable to MUS. However, the noteworthy disadvantages of Burch colposuspension include a high rate of urinary retention. This increased risk of urinary retention is due to the acute angle of the stitches, and is a problem that Burch colposuspension shares with the retropubic sling, a type of acutely-angled MUS. A variant of the retropubic sling, the transobturator tape (TOT), has shown that a rounder angle of elevation significantly reduces the risk of urinary retention. As such, this study proposes a novel technique of laparoscopic obturator urethropexy (LOU) as an alternative to the traditional Burch colposuspension.

In this new proposed technique, stitches are placed into the obturator internus fascia rather than Cooper's ligament, reducing the angle of elevation of the bladder neck, aiming to lower the risk of post-operative urinary retention. The aim of our randomized control trial is to assess the effectiveness of LOU compared to Burch colposuspension in terms of urinary continence. Our secondary aim is to report on perioperative and postoperative complications, functional outcomes including urinary retention, recurrent urinary tract infection, recurrent/persistent urgency, de novo urgency, recurrent SUI, and sexual function, as well as overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and be able to read and write English
* Women with symptomatic SUI, stress predominant mixed urinary incontinence symptoms confirmed on urodynamic study (UDS), or occult SUI (i.e. demonstrable urinary leakage on preoperative urodynamics with prolapse reduction in a patient without overt urinary incontinence symptoms), including women undergoing concomitant pelvic organ prolapse (POP) surgery or MUS sling removal

Exclusion Criteria:

* Known or suspected disease that affects bladder function (e.g. multiple sclerosis, Parkinson disease), including a known diagnosis of voiding dysfunction
* Pregnancy
* Desired fertility
* Urethral diverticulum
* History of radical pelvic surgery or pelvic radiation therapy
* Current chemotherapy or radiation therapy for malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Continence Rates | 1 year
  Patient reported symptoms of incontinence

SECONDARY OUTCOMES:
Objective continence rates | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Objective continence rates will be assessed with a cough test and a one-hour pad test.
Perioperative and postoperative complications | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Perioperative and postoperative complications will be assessed using the Clavien-Dindo (CD) classification.
Urinary retention | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Urinary retention will be assessed by an elevated post-void residual urine
Recurrent urinary tract infection | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Recurrent urinary tract infection will be assessed through a urine culture
Recurrent/persistent/de novo urgency | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Recurrent/persistent/de novo urgency will be based on patient symptoms
Recurrent SUI | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Recurrent SUI will be assessed through a cough test/a one-hour pad test
Sexual function | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Using the Female Sexual Function Index-6 (FSFI-6).
Overall quality of life | 6 weeks, 3 months, 6 months, 1 year and yearly up to 10 years
  Using the Pelvic Floor Distress Inventory-20 (PFDI-20).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.